CLINICAL TRIAL: NCT01949337
Title: Phase III Trial of Enzalutamide (NSC# 766085) Versus Enzalutamide, Abiraterone and Prednisone for Castration Resistant Metastatic Prostate Cancer
Brief Title: Enzalutamide With or Without Abiraterone and Prednisone in Treating Patients With Castration-Resistant Metastatic Prostate Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Astellas Pharma US, Inc. (Industry); Medivation, Inc. (Industry); Biologics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A031201; U10CA031946 (NIH); NCI-2013-01737 (Registry Identifier: Clinical Trial Reporting Program)
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Results first posted 2020-06-01 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Adenocarcinoma of the Prostate; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; abiraterone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: (enzalutamide) (Experimental): Patients receive enzalutamide 160 mg PO QD. Treatment will continue until confirmed disease progression or unacceptable toxicity.
  Interventions: Drug: enzalutamide
- Arm B: (enzalutamide, abiraterone, prednisone) (Experimental): Patients receive enzalutamide 160 mg PO QD, abiraterone 1000 mg PO QD, and prednisone 5 mg PO BID. Treatment will continue until confirmed disease progression or unacceptable toxicity.
  Interventions: Drug: enzalutamide; Drug: abiraterone; Drug: prednisone

INTERVENTIONS:
Drug: enzalutamide — Enzalutamide 160 mg daily, orally
Drug: abiraterone — abiraterone 1000 mg daily, orally
  Arms: Arm B: (enzalutamide, abiraterone, prednisone)
Drug: prednisone — prednisone 5 mg twice daily, orally
  Arms: Arm B: (enzalutamide, abiraterone, prednisone)

SUMMARY:
This randomized phase III trial studies enzalutamide to see how well it works compared to enzalutamide, abiraterone, and prednisone in treating patients with castration-resistant metastatic prostate cancer. Androgens can cause the growth of prostate cancer cells. Drugs, such as enzalutamide, abiraterone acetate, and prednisone, may lessen the amount of androgens made by the body.

DETAILED DESCRIPTION:
Patients are randomized to one of two treatment groups: enzalutamide or enzalutamide, abiraterone and prednisone. Treatment will continue until disease progression or unacceptable toxicity. Patients are followed for clinical outcomes for a maximum of 5 years post study treatment. The primary and secondary objectives are described below.

1. Primary Objective:

   To compare the overall survival of patients with progressive metastatic castration-resistant prostate cancer (CRPC) treated with either enzalutamide only or enzalutamide with abiraterone and prednisone
2. Secondary Objectives:

   * To assess the grade 3 or higher toxicity profile and compare safety by treatment arm.
   * To assess and compare post-treatment prostate-specific antigen (PSA) declines by treatment arm.
   * To compare radiographic progression free survival defined by Prostate Cancer Working Group 2 (PCWG2), and objective response rate, by treatment arm.
   * To test for radiographic progression free survival (rPFS) treatment interaction in predicting overall survival.
   * To assess pre- and post-treatment measures of tumor burden and bone activity using sodium fluoride (NaF) positron emission tomography (PET)/computed tomography (CT) and technetium (Tc) methylene diphosphonate (MDP) bone scintigraphy and correlate these measures with overall survival.
   * To develop and validate prognostic and predictive models of overall survival that include baseline clinical and molecular markers.

ELIGIBILITY:
Eligibility Criteria:

1. Documentation of Disease - Progressive castration-resistant metastatic prostate cancer with histologically or cytologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features
2. Patients must have measurable or non-measurable disease:

   1. Measurable Disease - For visceral or extra nodal lesions to be considered measurable, they must be ≥ 10 mm in one dimension, using spiral CT. For lymph nodes to be considered measurable (ie, target or evaluable lesions), they must be ≥ 20 mm in at least one dimension, using spiral CT.
   2. Non-Measurable Disease - All other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly non-measurable lesions. Lesions that are considered non-measurable include bone lesions (only).
   3. Patients with node only disease (ie, no presence of visceral, extra nodal lesions or bone lesions) must have node(s) that measure ≥ 15 mm in short axis.
3. Progressive Disease - Patients must have progressive disease at study entry defined as one or more of the following three criteria that occurred while the patient was on androgen deprivation therapy. For patients enrolling on the basis of soft tissue or bone progression, the baseline scan must show progression relative to a comparison scan. If the comparison scan is not available, the baseline scan report must reference the previous scan to document progression.

   1. PSA progression defined by a minimum of two rising PSA levels with an interval of ≥ 1 week between each determination. Patients who received an anti-androgen must have progression documented by a minimum of two rising PSA levels with an interval of ≥ 1 week between each determination such that at least the second of these rises is ≥ 4 weeks since last flutamide, bicalutamide or nilutamide.

      The PSA value at the screening should be ≥ 2 µg/L (2 ng/mL) .
   2. Soft tissue disease progression defined by the protocol
   3. Bone disease progression defined by the Prostate Cancer Working Group 2 (PCWG2) with two or more new lesions on bone scan
4. Prior Treatment

   1. No treatment with prior taxane-based chemotherapy for metastatic disease

      * Patients who received prior taxane-based chemotherapy as neoadjuvant or adjuvant therapy for local disease, or who received taxane-based therapy in the PSA clinical (non-metastatic) state is allowable provided that the total duration of exposure was six cycles or less and chemotherapy was completed more than 6 months prior to registration
      * Taxane-based chemotherapy that was aborted due to allergic reactions or intolerance to chemotherapy and therefore received one cycle of prior therapy is allowable
   2. No prior enzalutamide, abiraterone or other novel antiandrogen or androgen synthesis inhibitor
   3. No treatment with any of the following for prostate cancer within 4 weeks prior to enrollment:

      * Hormonal therapy (e.g., androgen receptor [AR] antagonists, 5 alpha reductase inhibitors, estrogens) Note: Treatment with bicalutamide and nilutamide within 4 weeks prior to enrollment is not allowed. Treatment with flutamide within 4 weeks prior to enrollment is not allowed. Treatment with all other gonadotropin- releasing hormone (GnRH) analogues or antagonists is allowed.
      * Chemotherapy
      * Biologic therapy
      * Investigational therapy
      * Immunotherapy
   4. No use of herbal products that may decrease PSA levels within 4 weeks prior to enrollment
   5. No use of systemic steroids greater than the equivalent of 10 mg of prednisone/prednisolone per day within 4 weeks prior to enrollment
   6. No prior use of ketoconazole for greater than 7 days
   7. No prior radiation therapy or radionuclide therapy for the treatment of metastasis within four weeks prior to enrollment
   8. Patients receiving bisphosphonate therapy or denosumab must have been on a stable dose for at least 4 weeks prior to enrollment
   9. Patients must maintain ongoing androgen deprivation therapy with a GnRH analogue, antagonist, or bilateral orchiectomy (i.e., surgical or medical castration)
5. Patient History

   1. No known or suspected brain metastases (NOTE: patients with treated epidural disease are allowed)
   2. No planned palliative procedures for alleviation of bone pain such as radiation therapy or surgery
   3. No structurally unstable bone lesions suggesting impending fracture
   4. No history of seizure or any condition that may increase the patient's seizure risk (e.g., prior cortical stroke, significant brain trauma). No history of transient ischemic attack (TIA) within 12 months of enrollment
   5. No clinically significant cardiovascular disease including:

      * Myocardial infarction (MI) within 6 months
      * Uncontrolled angina within 3 months
      * Congestive heart failure (CHF) with New York Heart Association (NYHA) class 3 or 4, or patients with NYHA class 3 or 4 in the past, unless a screening echocardiogram (echo) or multigated acquisition scan (MUGA) performed within three months demonstrates an ejection fraction (EF) > 45%
      * History of clinically significant ventricular arrhythmias (e.g., ventricular tachycardia, ventricular fibrillation, torsades de pointes)
      * History of Mobitz II second degree or third degree heart block without a permanent pacemaker in place
      * Hypotension (systolic blood pressure [BP] < 86 mmHg) or bradycardia (< 50 bpm) at screening
      * Uncontrolled hypertension (systolic BP > 170 mmHg or diastolic BP > 105 mmHg at screening)
   6. No gastrointestinal (GI) disorder that negatively affects absorption
   7. No major surgery within 4 weeks prior to enrollment
6. Age and performance status

   1. Age ≥ 18 years of age
   2. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
   3. Asymptomatic or mildly symptomatic from prostate cancer
7. Required Initial Laboratory Values

   1. Granulocytes ≥ 1,500/µL
   2. Platelet count ≥ 100,000/µL
   3. Hemoglobin ≥ 9 g/dL
   4. Creatinine ≤ 2 x upper limits of normal (ULN)
   5. Bilirubin ≤ 1.5 x ULN
   6. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 2 x ULN
   7. Albumin ≥ 3 g/dl
   8. Total testosterone ≤ 50 ng/dL (1.7 nmol/L)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1311 (Actual)
Dates: Start 2014-01-22 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2024-08-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, M.D., Study Chair — Memorial Sloan Kettering Cancer Center
Locations (539):
- United States (527):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Southern Cancer Center PC-Providence, Mobile, Alabama
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veteran's Administration Medical Center, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Hospital, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - University Oncology Associates, Fresno, California
  - California Cancer Center - North Fresno, Fresno, California
  - Kaiser Permanente, Fresno, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Feather River Cancer Center, Paradise, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Sharp Memorial Hospital, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - Veterans Administration-San Diego Medical Center, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Saint Joseph's Medical Center, Stockton, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - The Shaw Regional Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Greenwich Hospital, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Veterans Affairs Medical Center -Washington DC, Washington D.C., District of Columbia
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Northside Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Hawaii Oncology Inc-POB I, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Hines Veterans Administration Hospital, Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Quincy Medical Group-Clinic, Quincy, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc - Jefferson Boulevard, Fort Wayne, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - The Community Hospital, Munster, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Hematology Oncology Associates-Quad Cities, Bettendorf, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Iowa City VA Healthcare System, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Medical Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Montgomery General Hospital-Olney, Olney, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis Veterans Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - The West Clinic - Corinth, Corinth, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Barnes-Jewish West County Hospital, Creve Coeur, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-North, Kansas City, Missouri
  - The University of Kansas Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Saint Joseph Hospital, Nashua, New Hampshire
  - Norris Cotton Cancer Center-Nashua, Nashua, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Memorial Sloan Kettering Cancer Center at Basking Ridge, Basking Ridge, New Jersey
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Virtua Memorial, Mount Holly, New Jersey
  - The Valley Hospital-Luckow Pavilion, Paramus, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Kings County Hospital, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Veterans Affairs Western New York Health Care System-Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center Commack, Commack, New York
  - Arnot Ogden Medical Center/Falck Cancer Center, Elmira, New York
  - Memorial Sloan-Kettering Cancer Center West Harrison, Harrison, New York
  - North Shore-LIJ Health System/Center for Advanced Medicine, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - University of Rochester, Rochester, New York
  - Memorial Sloan Kettering Cancer Center Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Cancer Center Sleepy Hollow, Sleepy Hollow, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Syracuse Veterans Administration Medical Center, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Bronx Veterans Administration Medical Center, The Bronx, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Oncology Specialists of Charlotte, Charlotte, North Carolina
  - Southern Oncology Specialists-Charlotte, Charlotte, North Carolina
  - Durham Veterans Affairs Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Lake Norman Hematology Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Southern Oncology Specialists-Huntersville, Huntersville, North Carolina
  - Novant Health Oncology Specialists-Kernersville, Kernersville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Novant Health Cancer Specialists-Matthews, Matthews, North Carolina
  - Lake Norman Hematology Oncology Specialists-Mooresville, Mooresville, North Carolina
  - Novant Health Oncology Specialists-Mount Airy, Mount Airy, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Carolina Oncology Associates PA, Salisbury, North Carolina
  - Veterans Administration Medical Center, Salisbury, North Carolina
  - Novant Health Oncology Specialists-Statesville, Statesville, North Carolina
  - Novant Health Oncology Specialists-Davidson County, Thomasville, North Carolina
  - Marion L Shepard Cancer Center at Vidant Beaufort Hospital, Washington, North Carolina
  - Novant Health Oncology Specialists-Wilkesboro, Wilkesboro, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Novant Health Oncology Specialists, Winston-Salem, North Carolina
  - Winston-Salem Health Care, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Summa Barberton Hospital, Barberton, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Geaugra Hospital, Chardon, Ohio
  - University of Cincinnati/Barrett Cancer Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Ireland Cancer Center Landerbrook Health Center, Mayfield Heights, Ohio
  - Summa Health Center at Lake Medina, Medina, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center Ireland Cancer Center, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Ireland Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - University Pointe, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH-Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Good Samaritan Hospital, Corvallis, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Saint Mary Medical and Regional Cancer Center, Langhorne, Pennsylvania
  - Allegheny Valley Hospital, Natrona Heights, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Roger Williams Medical Center, Providence, Rhode Island
  - Roper Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates-Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Hematology Oncology Associates PA-St. Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - The West Clinic - Wolf River, Germantown, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Vermont College of Medicine, Burlington, Vermont
  - White River Junction Veteran Administration Medical Center, White River Junction, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Memorial Hospital Of Martinsville, Martinsville, Virginia
  - Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Shenandoah Oncology Associates PC, Winchester, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Saint Agnes Hospital/Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercy Health System, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - William S Middleton VA Medical Center, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Wheaton Franciscan Cancer Care - All Saints, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
- Canada (9):
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - The Moncton Hospital, Moncton, New Brunswick
  - The Vitalite Health Network - Dr Leon Richard Oncology Centre, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Cambridge Memorial Hospital, Cambridge, Ontario
  - Grand River Regional Cancer Centre at Grand River Hospital, Kitchener, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Puerto Rico (3):
  - San Juan Veterans Affairs Medical Center, San Juan
  - Fundacion De Investigacion de Diego, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Derived] Norton N, Larson NB, Jenkins GD, Beumer JH, Langevin B, Gobbaru J, Morris MJ, Nakamura Y, Kroetz DL, Zhu HJ, O'Donnell PH, Lewis LD, Hertz DL. Association of SULT2A1 Locus With Abiraterone Clearance in the Alliance A031201: Randomized Phase III Study of Enzalutamide Compared With Enzalutamide Plus Abiraterone for Metastatic Castration-Resistant Prostate Cancer. Clin Transl Sci. 2025 Dec;18(12):e70425. doi: 10.1111/cts.70425. PMID 41346252
- [Derived] Knutson TP, Luo B, Kobilka A, Lyman J, Guo S, Munro SA, Li Y, Heer R, Gaughan L, Morris MJ, Beltran H, Ryan CJ, Antonarakis ES, Armstrong AJ, Halabi S, Dehm SM. AR alterations inform circulating tumor DNA detection in metastatic castration resistant prostate cancer patients. Nat Commun. 2024 Dec 11;15(1):10648. doi: 10.1038/s41467-024-54847-1. PMID 39663356
- [Derived] Morris MJ, Heller G, Hillman DW, Bobek O, Ryan C, Antonarakis ES, Bryce AH, Hahn O, Beltran H, Armstrong AJ, Schwartz L, Lewis LD, Beumer JH, Langevin B, McGary EC, Mehan PT, Goldkorn A, Roth BJ, Xiao H, Watt C, Taplin ME, Halabi S, Small EJ. Randomized Phase III Study of Enzalutamide Compared With Enzalutamide Plus Abiraterone for Metastatic Castration-Resistant Prostate Cancer (Alliance A031201 Trial). J Clin Oncol. 2023 Jun 20;41(18):3352-3362. doi: 10.1200/JCO.22.02394. Epub 2023 Mar 30. PMID 36996380

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: (Enzalutamide) | Arm B: (Enzalutamide, Abiraterone, Prednisone)
Started | 657 | 654
Completed | 657 | 654
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: (Enzalutamide) | Arm B: (Enzalutamide, Abiraterone, Prednisone) | Total
Number analyzed (Participants) | 657 | 654 | 1311
Age, Customized [Count of Participants; unit: Participants]
  Age categories: < 60 years | 53 | 66 | 119
  Age categories: 60-69 years | 198 | 193 | 391
  Age categories: 70-79 years | 238 | 226 | 464
  Age categories: 80+ years | 168 | 169 | 337
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 657 | 654 | 1311
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 14 | 14 | 28
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 84 | 78 | 162
  White | 543 | 545 | 1088
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 13 | 27
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 376 | 387 | 763
    1 | 280 | 267 | 547
    Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from study registration to death due to any cause.
Time Frame: Up to 5 years post treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: (Enzalutamide) | Arm B: (Enzalutamide, Abiraterone, Prednisone)
Number analyzed (Participants) | 657 | 654
months | 32.5 [30.4 to 35.4] | 34.2 [31.8 to 37.5]
Statistical Analysis 1: Comparison: Arm A: (Enzalutamide) vs Arm B: (Enzalutamide, Abiraterone, Prednisone); Test type: Superiority; p = 0.33, Log Rank; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.80 to 1.08]

2. Secondary Outcome: Number of Participants Who Has Experienced at Least One Toxicity (Defined as a Grade 3 or Higher Adverse Event Deemed at Least Possibly Related to Treatment)
Description: The number of participants who has experienced at least one toxicity (defined as a grade 3 or higher adverse event deemed at least possibly related to treatment)
Time Frame: Up to 5 years post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: (Enzalutamide) | Arm B: (Enzalutamide, Abiraterone, Prednisone)
Number analyzed (Participants) | 657 | 654
Participants | 167 | 287

3. Secondary Outcome: Decline in Prostate Specific Antigen (PSA)
Time Frame: Up to 5 years post treatment
Reporting Status: Not Posted, anticipated posting 2023-08

4. Secondary Outcome: Progression Free Survival (PFS)
Time Frame: Up to 5 years post treatment
Reporting Status: Not Posted, anticipated posting 2023-08

5. Secondary Outcome: Objective Response Rate
Time Frame: Up to 5 years post treatment
Reporting Status: Not Posted, anticipated posting 2023-08

6. Secondary Outcome: Radiographic Progression Free Survival (rPFS)
Time Frame: Up to 5 years post treatment
Reporting Status: Not Posted, anticipated posting 2023-08

7. Secondary Outcome: Tumor Burden and Bone Activity
Time Frame: Up to 5 years post treatment
Reporting Status: Not Posted, anticipated posting 2023-08

ADVERSE EVENTS:
Time Frame: Up to 5 years post treatment
Arm/Group | Arm A: (Enzalutamide) | Arm B: (Enzalutamide, Abiraterone, Prednisone)
All-Cause Mortality (participants affected / at risk) | 372/657 | 339/654
Serious Adverse Events (participants affected / at risk) | 232/657 | 269/654
Other Adverse Events (participants affected / at risk) | 645/657 | 627/654
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: (Enzalutamide) (N=657) | Arm B: (Enzalutamide, Abiraterone, Prednisone) (N=654)
Anemia (Blood and lymphatic system disorders) | 11 (12) | 8 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 4 (4) | 1 (1)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 12 (14)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 8 (8) | 7 (10)
Chest pain - cardiac (Cardiac disorders) | 7 (9) | 7 (10)
Heart failure (Cardiac disorders) | 3 (4) | 6 (8)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 7 (7) | 6 (6)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (3)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (11) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 5 (7)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (2)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (2) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 1 (3)
Constipation (Gastrointestinal disorders) | 7 (9) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 5 (5)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (6) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 4 (5)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (11) | 10 (11)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 2 (4)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Visceral arterial ischemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 6 (8) | 7 (7)
Chills (General disorders) | 2 (2) | 3 (3)
Death NOS (General disorders) | 2 (2) | 5 (5)
Edema limbs (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 24 (32) | 28 (34)
Fever (General disorders) | 3 (3) | 8 (8)
Flu like symptoms (General disorders) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 1 (1) | 2 (2)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1) | 4 (4)
Localized edema (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 5 (6)
Pain (General disorders) | 3 (3) | 2 (2)
Sudden death NOS (General disorders) | 1 (1) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Anaphylaxis (Immune system disorders) | 0 (0) | 1 (2)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1)
Bone infection (Infections and infestations) | 0 (0) | 2 (3)
Bronchial infection (Infections and infestations) | 2 (2) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 2 (2)
Infections and infestations - Oth spec (Infections and infestations) | 4 (6) | 7 (8)
Joint infection (Infections and infestations) | 1 (1) | 1 (1)
Lung infection (Infections and infestations) | 4 (4) | 11 (11)
Sepsis (Infections and infestations) | 6 (6) | 16 (23)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 3 (3)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (6) | 0 (0)
Urinary tract infection (Infections and infestations) | 9 (11) | 26 (37)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aortic injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 16 (18) | 12 (14)
Fracture (Injury, poisoning and procedural complications) | 5 (6) | 9 (10)
Hip fracture (Injury, poisoning and procedural complications) | 6 (8) | 6 (7)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 5 (6) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 19 (29)
Alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 14 (20)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (3)
CPK increased (Investigations) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 3 (3) | 3 (4)
Ejection fraction decreased (Investigations) | 0 (0) | 2 (2)
INR increased (Investigations) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 2 (2) | 3 (3)
Lipase increased (Investigations) | 0 (0) | 2 (3)
Lymphocyte count decreased (Investigations) | 6 (6) | 3 (4)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (3)
Weight loss (Investigations) | 5 (7) | 2 (2)
White blood cell decreased (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 4 (5) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 7 (8) | 12 (13)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (8) | 5 (5)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 13 (14)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 7 (7) | 5 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 6 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 13 (15) | 8 (10)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 (8) | 18 (22)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 9 (12)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 5 (5) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 (19) | 27 (38)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Amnesia (Nervous system disorders) | 2 (2) | 0 (0)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6) | 8 (10)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 3 (4)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (7) | 5 (6)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 3 (3) | 3 (3)
Nervous system disorders - Oth spec (Nervous system disorders) | 3 (3) | 4 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Radiculitis (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 3 (3)
Stroke (Nervous system disorders) | 9 (10) | 8 (9)
Syncope (Nervous system disorders) | 7 (7) | 6 (6)
Transient ischemic attacks (Nervous system disorders) | 1 (2) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Confusion (Psychiatric disorders) | 5 (5) | 8 (9)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (7) | 1 (1)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 10 (11)
Bladder perforation (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 2 (4)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 10 (10) | 10 (10)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 5 (5) | 4 (4)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 4 (5)
Urinary tract obstruction (Renal and urinary disorders) | 5 (5) | 6 (6)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 15 (19) | 15 (17)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Social circumstances - Other, specify (Social circumstances) | 1 (1) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 7 (14) | 1 (1)
Hematoma (Vascular disorders) | 1 (3) | 2 (2)
Hot flashes (Vascular disorders) | 11 (18) | 8 (10)
Hypertension (Vascular disorders) | 26 (39) | 31 (44)
Hypotension (Vascular disorders) | 3 (3) | 5 (5)
Peripheral ischemia (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 10 (13) | 3 (3)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: (Enzalutamide) (N=657) | Arm B: (Enzalutamide, Abiraterone, Prednisone) (N=654)
Anemia (Blood and lymphatic system disorders) | 188 (1185) | 170 (1064)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 5 (10) | 9 (38)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (2) | 1 (2)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (7)
Atrial fibrillation (Cardiac disorders) | 5 (33) | 7 (21)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 3 (6) | 7 (20)
Chest pain - cardiac (Cardiac disorders) | 4 (5) | 8 (9)
Heart failure (Cardiac disorders) | 1 (1) | 3 (3)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 6 (10) | 5 (14)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 6 (21) | 9 (40)
Sinus tachycardia (Cardiac disorders) | 4 (5) | 5 (15)
Supraventricular tachycardia (Cardiac disorders) | 1 (2) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Congen, family, genetic disord -Oth spec (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 1 (2) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 2 (5)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 6 (26) | 6 (23)
Tinnitus (Ear and labyrinth disorders) | 9 (33) | 10 (32)
Vertigo (Ear and labyrinth disorders) | 7 (43) | 7 (27)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 2 (6)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (20) | 0 (0)
Blurred vision (Eye disorders) | 15 (76) | 18 (38)
Cataract (Eye disorders) | 2 (2) | 4 (15)
Dry eye (Eye disorders) | 3 (7) | 2 (15)
Eye disorders - Other, specify (Eye disorders) | 10 (23) | 10 (40)
Eye pain (Eye disorders) | 1 (1) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 1 (3)
Glaucoma (Eye disorders) | 1 (1) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 1 (3)
Watering eyes (Eye disorders) | 3 (19) | 2 (26)
Abdominal distension (Gastrointestinal disorders) | 5 (13) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 28 (88) | 22 (76)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 8 (14) | 6 (31)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 1 (10) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 245 (1509) | 216 (1315)
Dental caries (Gastrointestinal disorders) | 1 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 201 (1016) | 172 (530)
Dry mouth (Gastrointestinal disorders) | 13 (91) | 11 (58)
Dyspepsia (Gastrointestinal disorders) | 129 (682) | 132 (678)
Dysphagia (Gastrointestinal disorders) | 9 (30) | 5 (6)
Esophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 1 (1) | 3 (4)
Flatulence (Gastrointestinal disorders) | 12 (129) | 2 (4)
Gastritis (Gastrointestinal disorders) | 2 (4) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 10 (44) | 12 (38)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 12 (20) | 13 (47)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (5)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 4 (32) | 2 (8)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (3) | 2 (5)
Nausea (Gastrointestinal disorders) | 96 (288) | 120 (384)
Oral dysesthesia (Gastrointestinal disorders) | 2 (4) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (2) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (10) | 2 (2)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 2 (3)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 6 (14) | 1 (3)
Tooth development disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth discoloration (Gastrointestinal disorders) | 0 (0) | 1 (15)
Toothache (Gastrointestinal disorders) | 2 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 87 (165) | 80 (133)
Chills (General disorders) | 6 (6) | 7 (11)
Edema face (General disorders) | 1 (1) | 5 (36)
Edema limbs (General disorders) | 173 (1354) | 196 (1407)
Facial pain (General disorders) | 1 (1) | 1 (5)
Fatigue (General disorders) | 556 (7352) | 526 (6588)
Fever (General disorders) | 5 (7) | 6 (7)
Flu like symptoms (General disorders) | 12 (15) | 8 (11)
Gait disturbance (General disorders) | 9 (63) | 10 (32)
Gen disord and admin site conds-Oth spec (General disorders) | 14 (26) | 16 (20)
Injection site reaction (General disorders) | 1 (2) | 1 (1)
Localized edema (General disorders) | 5 (23) | 6 (13)
Malaise (General disorders) | 6 (26) | 3 (7)
Neck edema (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 13 (23) | 5 (6)
Pain (General disorders) | 44 (150) | 43 (199)
Bile duct stenosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 4 (4)
Allergic reaction (Immune system disorders) | 2 (3) | 2 (4)
Anorectal infection (Infections and infestations) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1) | 4 (9)
Bronchial infection (Infections and infestations) | 5 (5) | 1 (1)
Conjunctivitis (Infections and infestations) | 5 (13) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 1 (1)
Gum infection (Infections and infestations) | 3 (3) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 11 (18) | 20 (23)
Joint infection (Infections and infestations) | 1 (2) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (2)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 2 (2) | 1 (2)
Lung infection (Infections and infestations) | 1 (1) | 2 (2)
Mucosal infection (Infections and infestations) | 2 (2) | 4 (8)
Nail infection (Infections and infestations) | 2 (2) | 2 (2)
Otitis media (Infections and infestations) | 1 (1) | 2 (3)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (5)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Scrotal infection (Infections and infestations) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 3 (3)
Sinusitis (Infections and infestations) | 2 (2) | 4 (6)
Skin infection (Infections and infestations) | 7 (9) | 10 (14)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 3 (3) | 2 (2)
Upper respiratory infection (Infections and infestations) | 18 (23) | 13 (15)
Urinary tract infection (Infections and infestations) | 16 (20) | 22 (37)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Aortic injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 12 (38) | 30 (137)
Fall (Injury, poisoning and procedural complications) | 31 (43) | 38 (66)
Fracture (Injury, poisoning and procedural complications) | 6 (21) | 9 (37)
Hip fracture (Injury, poisoning and procedural complications) | 2 (3) | 1 (1)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 5 (10) | 3 (5)
Intraoperative head and neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 6 (18)
Urostomy obstruction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (4) | 1 (8)
Alanine aminotransferase increased (Investigations) | 40 (99) | 215 (703)
Alkaline phosphatase increased (Investigations) | 66 (210) | 88 (281)
Aspartate aminotransferase increased (Investigations) | 73 (232) | 217 (729)
Blood antidiuretic hormone abnormal (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 44 (154) | 87 (328)
CO diffusing capacity decreased (Investigations) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 2 (2) | 1 (1)
Cholesterol high (Investigations) | 7 (41) | 6 (55)
Creatinine increased (Investigations) | 45 (190) | 35 (103)
GGT increased (Investigations) | 1 (1) | 0 (0)
Hemoglobin increased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 2 (2) | 2 (3)
Investigations - Other, specify (Investigations) | 11 (22) | 14 (44)
Lipase increased (Investigations) | 1 (1) | 1 (1)
Lymphocyte count decreased (Investigations) | 56 (259) | 67 (300)
Lymphocyte count increased (Investigations) | 2 (3) | 2 (2)
Neutrophil count decreased (Investigations) | 33 (173) | 14 (66)
Platelet count decreased (Investigations) | 38 (175) | 41 (202)
Weight gain (Investigations) | 15 (93) | 10 (62)
Weight loss (Investigations) | 60 (222) | 72 (295)
White blood cell decreased (Investigations) | 65 (451) | 36 (103)
Anorexia (Metabolism and nutrition disorders) | 85 (458) | 86 (301)
Dehydration (Metabolism and nutrition disorders) | 8 (9) | 6 (9)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 3 (59)
Hypercalcemia (Metabolism and nutrition disorders) | 18 (30) | 16 (29)
Hyperglycemia (Metabolism and nutrition disorders) | 338 (2782) | 321 (2468)
Hyperkalemia (Metabolism and nutrition disorders) | 32 (80) | 15 (68)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 18 (35) | 22 (30)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 7 (32) | 6 (8)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 50 (165) | 58 (189)
Hypocalcemia (Metabolism and nutrition disorders) | 27 (53) | 23 (53)
Hypoglycemia (Metabolism and nutrition disorders) | 7 (10) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 86 (220) | 179 (469)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (6) | 2 (11)
Hyponatremia (Metabolism and nutrition disorders) | 52 (136) | 47 (112)
Hypophosphatemia (Metabolism and nutrition disorders) | 11 (18) | 13 (29)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 8 (10) | 7 (39)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 291 (2233) | 227 (1798)
Arthritis (Musculoskeletal and connective tissue disorders) | 13 (30) | 14 (50)
Back pain (Musculoskeletal and connective tissue disorders) | 75 (260) | 65 (333)
Bone pain (Musculoskeletal and connective tissue disorders) | 300 (1751) | 261 (1524)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (4) | 1 (22)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (6)
Flank pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (14)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 42 (194) | 51 (231)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 17 (110) | 30 (106)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (16)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 21 (67) | 22 (110)
Myalgia (Musculoskeletal and connective tissue disorders) | 189 (1102) | 170 (915)
Neck pain (Musculoskeletal and connective tissue disorders) | 13 (51) | 7 (30)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 (16) | 2 (15)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (7) | 4 (21)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 49 (167) | 44 (220)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Akathisia (Nervous system disorders) | 3 (21) | 2 (2)
Amnesia (Nervous system disorders) | 1 (1) | 3 (3)
Ataxia (Nervous system disorders) | 3 (6) | 4 (14)
Brachial plexopathy (Nervous system disorders) | 1 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 11 (81) | 12 (113)
Concentration impairment (Nervous system disorders) | 5 (26) | 7 (55)
Dizziness (Nervous system disorders) | 64 (237) | 82 (298)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1)
Dysesthesia (Nervous system disorders) | 3 (26) | 0 (0)
Dysgeusia (Nervous system disorders) | 42 (258) | 38 (161)
Dysphasia (Nervous system disorders) | 0 (0) | 2 (2)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (8)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 2 (2)
Facial nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 163 (1000) | 176 (826)
Lethargy (Nervous system disorders) | 2 (3) | 3 (9)
Memory impairment (Nervous system disorders) | 37 (255) | 39 (351)
Movements involuntary (Nervous system disorders) | 1 (3) | 2 (9)
Muscle weakness left-sided (Nervous system disorders) | 1 (1) | 2 (4)
Muscle weakness right-sided (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 13 (104) | 16 (88)
Neuralgia (Nervous system disorders) | 1 (2) | 2 (5)
Paresthesia (Nervous system disorders) | 12 (44) | 11 (44)
Peripheral motor neuropathy (Nervous system disorders) | 7 (36) | 8 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 43 (287) | 31 (123)
Presyncope (Nervous system disorders) | 2 (2) | 4 (4)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Spasticity (Nervous system disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 8 (8) | 5 (10)
Transient ischemic attacks (Nervous system disorders) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 8 (33) | 13 (60)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (2) | 5 (11)
Anxiety (Psychiatric disorders) | 27 (67) | 32 (182)
Confusion (Psychiatric disorders) | 15 (18) | 18 (51)
Delirium (Psychiatric disorders) | 1 (3) | 0 (0)
Depression (Psychiatric disorders) | 36 (155) | 44 (218)
Hallucinations (Psychiatric disorders) | 1 (1) | 1 (25)
Insomnia (Psychiatric disorders) | 210 (1574) | 203 (1503)
Irritability (Psychiatric disorders) | 4 (8) | 1 (1)
Libido decreased (Psychiatric disorders) | 2 (10) | 1 (3)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 3 (9) | 5 (9)
Restlessness (Psychiatric disorders) | 1 (10) | 3 (33)
Bladder spasm (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 7 (45) | 5 (30)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 2 (2)
Hematuria (Renal and urinary disorders) | 31 (69) | 31 (64)
Proteinuria (Renal and urinary disorders) | 0 (0) | 3 (14)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 21 (66) | 17 (51)
Renal calculi (Renal and urinary disorders) | 1 (1) | 3 (9)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 47 (243) | 44 (266)
Urinary incontinence (Renal and urinary disorders) | 26 (141) | 23 (136)
Urinary retention (Renal and urinary disorders) | 7 (16) | 13 (28)
Urinary tract obstruction (Renal and urinary disorders) | 3 (9) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 5 (12) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 12 (60) | 8 (27)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 2 (5)
Breast pain (Reproductive system and breast disorders) | 6 (28) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 21 (318) | 13 (184)
Genital edema (Reproductive system and breast disorders) | 1 (3) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 24 (243) | 5 (57)
Pelvic pain (Reproductive system and breast disorders) | 6 (9) | 6 (33)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (4)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 2 (3) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Testicular disorder (Reproductive system and breast disorders) | 1 (2) | 1 (3)
Testicular pain (Reproductive system and breast disorders) | 4 (13) | 6 (61)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 8 (77) | 16 (108)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 191 (899) | 206 (924)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 189 (1380) | 201 (1391)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 5 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 8 (33) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 14 (24) | 9 (48)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 3 (17) | 6 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 4 (18) | 4 (4)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 12 (17) | 2 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (9) | 12 (119)
Dry skin (Skin and subcutaneous tissue disorders) | 25 (146) | 16 (107)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 8 (52) | 6 (21)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 2 (29) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Nail ridging (Skin and subcutaneous tissue disorders) | 3 (14) | 2 (8)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 10 (46) | 14 (35)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (11) | 3 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 (62) | 22 (44)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 24 (98) | 26 (80)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (7) | 2 (8)
Social circumstances - Other, specify (Social circumstances) | 0 (0) | 1 (1)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 3 (4) | 3 (4)
Flushing (Vascular disorders) | 4 (34) | 10 (56)
Hematoma (Vascular disorders) | 5 (5) | 1 (1)
Hot flashes (Vascular disorders) | 416 (5649) | 438 (5781)
Hypertension (Vascular disorders) | 413 (5471) | 416 (5628)
Hypotension (Vascular disorders) | 11 (16) | 10 (11)
Lymph leakage (Vascular disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischemia (Vascular disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 4 (5)
Vascular disorders - Other, specify (Vascular disorders) | 5 (15) | 2 (31)
Vasculitis (Vascular disorders) | 1 (15) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT01949337/Prot_SAP_000.pdf